CLINICAL TRIAL: NCT07134166
Title: Observational Registry of Advanced Cardiac Imaging in Systemic Lupus Erythematosus and Other Inflammatory diseaseS
Brief Title: Cardiac Imaging in Systemic Disorders: the ORACLES Registry
Acronym: ORACLES
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP250892
Record Dates: First submitted 2025-06-26; First posted 2025-08-21 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-06

CONDITIONS: Lupus
Keywords: Cardiac imaging; cardiac magnetic resonance imaging,; cardiac computed tomography; coronary angiogram computed tomography; coronary artery calcium; epicardial adipose tissue; inflammation; systemic lupus erythematosus; sarcoidosis; vasculitis; histiocytosis; atherosclerosis; myocarditis; corticosteroids; cytokines
MeSH Terms: conditions — Inflammation; Lupus Erythematosus, Systemic; Sarcoidosis; Vasculitis; Histiocytosis; Atherosclerosis; Myocarditis | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: data collection — data collection

SUMMARY:
Autoimmune diseases affect a total of 5 to 10% of the population. These diseases are associated with an increased risk of developing cardiovascular pathologies. Modern cardiac imaging tools could provide a better understanding of these complications, enabling earlier diagnosis and detection of patients most at risk. Yet, the diagnostic and prognostic value of multimodal cardiac imaging in these diseases is under-researched. The current registry aimed at investigating the diagnostic and prognostic value of cardiac imaging in autoimmune and systemic disorders.

DETAILED DESCRIPTION:
This is an observational prospective registry including patients with systemic disorders and autoimmune diseases who benefit from cardiac imaging. This is a single-center registry (Hôpital Pitié-Salpêtrière). Collected data at baseline include clinical, biological and imaging data. The study is not interventional. It includes data generated from routine care. The main objective is the characterization of the cardiovascular phenotype of patients with autoimmune, systemic and/or inflammatory diseases. Secondary objectives include the development and validation of prognostic biomarkers, the identification and quantification of specific risk factors for cardiovascular disease, and the evaluation of tolerance and efficacy of conventional and innovative therapies

ELIGIBILITY:
Inclusion Criteria:

1. Suspected or diagnosed autoimmune, inflammatory and/or systemic disease.
2. Cross-sectional cardiac imaging including either nonenhanced cardiac computed tomography, enhanced coronary angiogram-computed tomography, or cardiac magnetic resonance imaging

Exclusion Criteria:

* Age < 18 years
* Objection to study participation
* Patient under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Suspected or diagnosed autoimmune, inflammatory and/or systemic disease.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2026-11 (Estimated); Primary Completion 2046-11 (Estimated); Study Completion 2046-11 (Estimated)

PRIMARY OUTCOMES:
MACE (major adverse cardiovascular events) | Through study completion, an average of 10 year
  Composite outcome of myocardial infarction, stroke or cardiovascular death.

SECONDARY OUTCOMES:
ASCVD (atherosclerotic cardiovascular disease) | Through study completion, an average of 10 year
  Composite outcome of acute coronary syndrome, stroke and peripheral artery disease.
Cardiovascular events (all) | Through study completion, an average of 10 year
  MACE, ASCVD, device implantation, coronary artery disease, heart failure, rhythm and conduction disorders, valvular disorders, cardiovascular interventions, fatal and non fatal.

IPD SHARING:
Plan to Share IPD: Yes
The procedures carried out with the French data privacy authority (CNIL, Commission nationale de l'informatique et des libertés) do not provide for the transmission of the database, nor do the information and consent documents signed by the patients.
  Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations.
Supporting Information: Study Protocol, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out of these time frame can also be submitted to the sponsor
Access Criteria: Researchers who provide a methodologically sound proposal